CLINICAL TRIAL: NCT00707798
Title: A Study to Evaluate GSK Biologicals' Candidate Formulations of Pneumococcal Vaccines (GSK2189242A) in Young Adults.
Brief Title: Evaluation of Pneumococcal Vaccine Formulations in Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111651
Record Dates: First submitted 2008-06-30; First posted 2008-07-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Young adults; Pneumococcal vaccine,; Streptococcus pneumoniae,
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (7):
- Formulation 1 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- Formulation 2 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- Formulation 3 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- Formulation 4 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- Formulation 5 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- Formulation 6 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A
- 23 valent pneumococcal vaccine (Active Comparator)
  Interventions: Biological: Pneumo 23™

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2189242A — Two doses of 0.5 ml will be administered intramuscularly; one dose at Month 0 and another at Month 2. Six different formulations of this vaccine will be tested
  Arms: Formulation 1; Formulation 2; Formulation 3; Formulation 4; Formulation 5; Formulation 6
Biological: Pneumo 23™ — One dose of 0.5 ml will be administered intramuscularly at Month 0, and a placebo dose to keep the blinding at Month 2
  Arms: 23 valent pneumococcal vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of pneumococcal vaccines in young adults. Subjects will be vaccinated twice with an interval of two months.

DETAILED DESCRIPTION:
This amendment was due to

* The addition of secondary endpoints for safety. The collection of data related to these secondary safety endpoints was already planned and the corresponding statistical analyses were described in the statistical section.
* The addition of an exclusion criterion regarding the administration of immunoglobulins and blood products. It is already included in the elimination criteria section. It impacts only immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female between, and including, 18 and 40 years old at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history, clinical examination and clinical laboratory assessment before entering into the study.
* If the subject is female, and of child-bearing potential, she agrees to use adequate contraception and not become pregnant for the duration of the study.

Exclusion Criteria:

* Previous vaccination against Streptococcus pneumoniae.
* Vaccination with diphtheria/tetanus toxoids within one month preceding the first dose of study vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period or participation to another pharmaceutical/vaccine study.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine, with the exception of the influenza vaccine which can be administered > 7 days preceding or > 7 days following each vaccine dose (after collection of 7-day safety data).
* Bacterial pneumonia within 3 years prior to 1st vaccination.
* Invasive pneumococcal disease (IPD) within 3 years prior to 1st vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of thrombocytopenia or bleeding disorder.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Current serious neurologic or mental disorders.
* Inflammatory processes such as known chronic active infections (e.g. Hepatitis B, C).
* All past or current malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders.
* Acute disease at the time of enrolment/vaccination.
* Physical examination positive for acrocyanosis, jaundice, splenomegaly.
* Acute or chronic, clinically significant anaemia, pulmonary, cardiovascular, hematologic , hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, at the discretion of the investigator.
* Laboratory evidence of haematological abnormalities.
* Laboratory evidence of biochemical abnormalities
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2009-01-15 (Actual); Study Completion 2009-01-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of any vaccine related and grade 3 solicited local and general adverse events | During a 7-day follow up period after each vaccine dose
Occurrence of any vaccine related and grade 3 unsolicited adverse events | During a 31-day follow up period after each vaccine dose
Occurrence of any vaccine related serious adverse events (SAE) | From Visit 1 to study conclusion
Occurrence of any grade 3 laboratory abnormalities | During a 7-day follow up period after each vaccine dose

SECONDARY OUTCOMES:
Occurrence of any solicited local and general adverse events | During a 7-day follow up period after each vaccine dose.
Occurrence of any unsolicited adverse events | During a 31-day follow up period after each vaccine dose
Occurrence of any haematological, biochemical, or urinary abnormalities | At 1 and 7 days after each vaccine dose
Anti-pneumococcal and anti-NTHi candidate vaccine antigens | At Days 0, 30 and 90

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Leroux-Roels G, Maes C, De Boever F, Traskine M, Ruggeberg JU, Borys D. Safety, reactogenicity and immunogenicity of a novel pneumococcal protein-based vaccine in adults: a phase I/II randomized clinical study. Vaccine. 2014 Nov 28;32(50):6838-46. doi: 10.1016/j.vaccine.2014.02.052. Epub 2014 Mar 6. PMID 24607003
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111651 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/111651?search=study&b%22b''%22#rs
- Available data/document: Informed Consent Form: 111651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register